CLINICAL TRIAL: NCT05662215
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CK-3828136 in Healthy Participants
Brief Title: A Single and Multiple Ascending Dose Study of CK-3828136 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early per sponsor decision.
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: CY 8011
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Healthy Participants
Keywords: CK-3828136, CK-136

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CK-3828136 for SAD Cohort (Experimental): Subjects will be assigned to one of approximately 8 planned dose cohorts and receive single doses of CK-3828136
  Interventions: Drug: CK-3828136
- Placebo for SAD Cohort (Placebo Comparator): Subjects will be assigned to one of approximately 8 planned cohorts and receive single doses of placebo
  Interventions: Drug: Placebo for CK-3828136
- CK-3828136 for MAD Cohort (Experimental): Subjects will be assigned to one of approximately 8 planned dose cohorts and receive multiple doses of CK-3828136
  Interventions: Drug: CK-3828136
- Placebo for MAD Cohort (Placebo Comparator): Subjects will be assigned to one of approximately 8 planned cohorts and receive single doses of placebo
  Interventions: Drug: Placebo for CK-3828136
- Food Effect (Experimental): Healthy subjects will be administered CK-3828136 with and without food in a cross-over fashion.
  Interventions: Drug: CK-3828136

INTERVENTIONS:
Drug: CK-3828136 — CK-3828136
  Arms: CK-3828136 for MAD Cohort; CK-3828136 for SAD Cohort; Food Effect
Drug: Placebo for CK-3828136 — Placebo for CK-3828136
  Arms: Placebo for MAD Cohort; Placebo for SAD Cohort

SUMMARY:
1. Learn about the safety and tolerability of CK-3828136 after a single dose and multiple doses in healthy subjects.
2. Find out how much CK-3828136 is in the blood after a single dose and multiple doses.
3. Determine the effect different doses of CK-3828136 on the pumping function of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged between 18 and 45 years (inclusive) with a body mass index between 18.0 and 30.0 kg/m2 (inclusive), with a body weight > 50.0 kg.

Exclusion Criteria:

Participants will not be enrolled in the study if they meet any of the following exclusion criteria at the screening visit, unless otherwise stated:

* History of any significant illness or disorder.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, hernia repair, and/or cholecystectomy will be allowed).
* History or presence of:

  1. additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).
  2. sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or clinically significant conduction abnormalities.
* Clinically significant illness within 4 weeks prior to check in.
* Participants with an inability to swallow tablets.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs | Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14; Time Frame for Food Effect Cohorts: Days 1 to 7 (Treatment Periods 1 and 2)
  To assess the safety and tolerability of CK-3828136 when administered orally as single or multiple doses to healthy participants

SECONDARY OUTCOMES:
Primary PK parameters of CK-3828136 including AUC | Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14; Time Frame for Food Effect Cohorts: Days 1 to 7 (Treatment Periods 1 and 2)
  To characterize the PK of CK-3828136 after single and multiple oral doses in healthy participants
Changes over time from baseline in echocardiographic parameters including, but not limited to, LVEF | Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14
  To characterize the PD effects of single and multiple oral doses of CK-3828136 in healthy participants Time Frame for SAD Cohorts: Day -1 - Day 7; Time Frame for MAD Cohorts: Day -1 - Day 14
PK parameters calculated using plasma CK-3828136 concentrations including AUC in fed and fasted state | Time Frame for Food Effect Cohort: Days 1 to 7 (Treatment Periods 1 and 2)
  PK parameters following single multiple doses in fed and fasted state

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics, MD, Study Director — Cytokinetics
Locations (1):
- Labcorp Clinical Research Unit Inc., Dallas, Texas, United States